CLINICAL TRIAL: NCT02774187
Title: Sorafenib Alone Versus Sorafenib Combined With Hepatic Arterial Chemoinfusion for Advanced HCC With Portal Vein Tumor Thrombosis: a Multicentre Randomised Controlled Trial
Brief Title: Sorafenib Alone Versus Sorafenib Combined With HAIC for Advanced HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Kaiping Central Hospital (Other); Guangzhou No.12 People's Hospital (Other Government); The First Affiliated Hospital of University of South China (Other)
Responsible Party: Principal Investigator, Shi Ming, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S021
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatic arterial infusion chemotherapy; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Folfox protocol; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib combined with HAIC (Experimental): Sorafenib combined with Hepatic arterial infusion chemotherapy with Folfox Protocol
  Interventions: Drug: Sorafenib; Procedure: Hepatic arterial infusion chemotherapy; Drug: Folfox Protocol
- Sorafenib alone (Active Comparator): Sorafenib alone
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — administration of Sorafenib
Procedure: Hepatic arterial infusion chemotherapy — administration of Oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
  Other Names: HAIC
  Arms: Sorafenib combined with HAIC
Drug: Folfox Protocol — Oxaliplatin , fluorouracil, and leucovorin
  Other Names: Oxaliplatin , fluorouracil, and leucovorin
  Arms: Sorafenib combined with HAIC

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sorafenib combined with hepatic arterial infusion chemotherapy (HAIC) compared with sorafenib Alone in patients with hepatocellular carcinoma (HCC) with major portal venous tumor thrombus (PVTT).

DETAILED DESCRIPTION:
The results of our preliminary pilot study suggested that sorafenib combined with hepatic arterial infusion chemotherapy (HAIC) may improve the survivals for advanced stage HCC. Thus, the investigators carried out this prospective randomized control study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* portal vein tumor thrumbus confirmed in two image techniques
* Eastern Cooperative Oncology Group performance status of 0 to 2
* with no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

  * Platelet count ≥ 75,000/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 30mmol/L
  * Serum albumin ≥ 30 g/L
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or PT/APTT within normal limits
  * Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 6 months
  Overall survival

SECONDARY OUTCOMES:
Time to progression | 6 months
  Time to progression
Adverse Events | 30 days
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v3.0
Number of of Patients developed Adverse Events | 30 days
  Number of of patients who developed adverse event. Postoperative adverse events were graded based on CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — The Department of Hepatobiliary Oncology of Sun Yat-sen University Cancer Center
Locations (5):
- China (5):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospita, Guangzhou, Guangdong
  - The Kaiping Center's Hospital, Kaiping, Guangdong
  - First Affiliated Hospital of University Of South China, Hengyang, Hunan

REFERENCES:
- [Result] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Result] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Result] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794
- [Result] Luo J, Guo RP, Lai EC, Zhang YJ, Lau WY, Chen MS, Shi M. Transarterial chemoembolization for unresectable hepatocellular carcinoma with portal vein tumor thrombosis: a prospective comparative study. Ann Surg Oncol. 2011 Feb;18(2):413-20. doi: 10.1245/s10434-010-1321-8. Epub 2010 Sep 14. PMID 20839057
- [Result] Ando E, Yamashita F, Tanaka M, Tanikawa K. A novel chemotherapy for advanced hepatocellular carcinoma with tumor thrombosis of the main trunk of the portal vein. Cancer. 1997 May 15;79(10):1890-6. doi: 10.1002/(sici)1097-0142(19970515)79:103.0.co;2-k. PMID 9149014
- [Result] Shi J, Lai EC, Li N, Guo WX, Xue J, Lau WY, Wu MC, Cheng SQ. A new classification for hepatocellular carcinoma with portal vein tumor thrombus. J Hepatobiliary Pancreat Sci. 2011 Jan;18(1):74-80. doi: 10.1007/s00534-010-0314-0. PMID 20686792
- [Result] Huang ZL, Luo J, Chen MS, Li JQ, Shi M. Blood neutrophil-to-lymphocyte ratio predicts survival in patients with unresectable hepatocellular carcinoma undergoing transarterial chemoembolization. J Vasc Interv Radiol. 2011 May;22(5):702-9. doi: 10.1016/j.jvir.2010.12.041. PMID 21514523
- [Result] Fan W, Zhang Y, Wang Y, Yao X, Yang J, Li J. Neutrophil-to-lymphocyte and platelet-to-lymphocyte ratios as predictors of survival and metastasis for recurrent hepatocellular carcinoma after transarterial chemoembolization. PLoS One. 2015 Mar 5;10(3):e0119312. doi: 10.1371/journal.pone.0119312. eCollection 2015. PMID 25742141
- [Derived] He M, Li Q, Zou R, Shen J, Fang W, Tan G, Zhou Y, Wu X, Xu L, Wei W, Le Y, Zhou Z, Zhao M, Guo Y, Guo R, Chen M, Shi M. Sorafenib Plus Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin vs Sorafenib Alone for Hepatocellular Carcinoma With Portal Vein Invasion: A Randomized Clinical Trial. JAMA Oncol. 2019 Jul 1;5(7):953-960. doi: 10.1001/jamaoncol.2019.0250. PMID 31070690